CLINICAL TRIAL: NCT03863197
Title: Treatment Algorithms Based on Muscle and Tendon Morphology - Progressive Supervised Home-based Strength Training in Children With Spastic Cerebral Palsy
Brief Title: Progressive Supervised Home-based Strength Training in Children With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other); University Ghent (Other); Queen Fabiola Children's University Hospital (Other)
Responsible Party: Principal Investigator, Kaat Desloovere, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: S59945
Record Dates: First submitted 2019-02-12; First posted 2019-03-05 (Actual); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Cerebral Palsy; Spastic Cerebral Palsy; Progressive Strength Training; Muscle morphology
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with waitlist control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): During a 12-week period children receive 3-4 sessions of progressive strength training per week on top of the usual care. All children will be provided with an individualized training program and supporting equipment. One or 2 session per week will be performed under supervision of the physical therapist, whilst the remaining sessions will be performed at home. Progression is closely monitored by the principal investigator and training programs are adjusted if necessary.
  Interventions: Behavioral: Progressive strength training
- Waitlist-control group (No Intervention): The waitlist-control group will continue their usual care without additional treatment for 12-weeks, followed by a 12-week period of progressive supervised home-based strength training.

INTERVENTIONS:
Behavioral: Progressive strength training — Progressive Supervised Home-based Strength Training
  Arms: Intervention group

SUMMARY:
A randomized controlled trail will be carried out to investigate the effect of a 12-week supervised home-based progressive strength intervention in children with spastic cerebral palsy aged 5-11 years. The results of this strength intervention aiming for increased strength and muscle hypertrophy will serve as input for a clinical decision making framework based on muscle and tendon architecture.

DETAILED DESCRIPTION:
Background: The alterations of morphological muscle and tendon properties are a primary determinant of the pathological muscle behaviour in spastic cerebral palsy (SCP). As treatments aim to reduce the progressive secondary problems, they are mainly directed at the muscle level. Muscle morphology features like volume, fascicle architecture and tendon properties are all responsive to treatment, but these treatment responses seem to be both patient and muscle-specific. Therefore, objective tools and protocols are needed for the evaluation of morphological muscle and tendon (MMT) properties in routine clinical practice. These are required to guide the patient-specific selection of appropriate, rationalized treatment choices and to determine the impact of these treatments on the MMT properties, the muscular impairment and function in children with SCP.

This intervention study is one out of three intervention studies focused on defining the effects of conservative treatments (strengthening, stretching and botulinum toxin injections) on muscle and tendon architecture. In this phase of the Treatment Algorithms based on Muscle and Tendon Morphology (TAMTA) project, we aim to develop specific guidelines for these treatment options linked to the MMT evaluation protocol. To achieve this goal, prediction models based on baseline MMT parameters for the prognosis of specific treatment outcomes will be developed from the data of the three intervention studies.

Aim: (1) determine whether the 12-week program of targeted progressive strengthening of the plantar flexors, the knee flexors and extensors leads to changes in the MMT properties of medial gastrocnemius, semitendinosus and rectus femoris, in the muscle strength and in gross motor function; and (2) determine the correlation between baseline MMT properties and the changes in the outcome parameters.

Methods/Design: A randomized controlled trial will be conducted in 40 ambulatory children with a confirmed diagnosis of SCP between 5 and 11 years of age. Participants will be randomized to the intervention group (who will additionally receive the strengthening program while continuing their usual care) or to the waitlist-control group (who will continue their usual care without additional treatment) using the randomization by minimization method (with influencing characteristics age and GMFCS level). Participants in the control group will be able to participate in the intervention after the control period. The MMT parameters of the medial gastrocnemius, tibialis anterior, semitendinosus and rectus femoris and the isometric and functional strength for the 4 related lower limb muscle groups (plantar flexors, dorsiflexors, knee flexors and knee extensors) as well as the gross motor function will be assessed before and after the 12-week program. After 6 weeks a short evaluation of the MMT parameters, isometric and functional strength will take place.

The change in primary outcome parameters before and after training of the intervention group will be compared to the data behaviour of the control group. Secondly, to explore the predictive value of specific baseline MMT parameters on treatment effect, both univariate and multivariate linear regression analyses will be conducted to identify significant predictive variables for the primary outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of SCP
* Aged 5-12 years
* GMFCS levels I-III (GMFCS = Gross Motor Function Classification Score, expressing the overall functional level of impairment)
* Sufficient cooperation to comprehend and complete the test procedure

Exclusion Criteria:

* Non-ambulatory
* Botulinum toxin A injections six months prior to enrollment
* Lower limb surgery two years prior to enrollment
* Presence of ataxia or dystonia
* Cognitive problems that impede measurements
* Severe co-morbidities (severe epilepsy, non-correctable visual impairment, autism spectrum disorders, mental problems that prevent comprehensiveness of the tasks)

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Desloovere, Dr, Study Director — KU Leuven
Locations (2):
- Belgium (2):
  - Universiteit Gent, Ghent
  - KU Leuven, Leuven

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hanssen B, Peeters N, Vandekerckhove I, De Beukelaer N, Bar-On L, Molenaers G, Van Campenhout A, Degelaen M, Van den Broeck C, Calders P, Desloovere K. The Contribution of Decreased Muscle Size to Muscle Weakness in Children With Spastic Cerebral Palsy. Front Neurol. 2021 Jul 26;12:692582. doi: 10.3389/fneur.2021.692582. eCollection 2021. PMID 34381414
- [Result] Hanssen B, Peeters N, De Beukelaer N, Vannerom A, Peeters L, Molenaers G, Van Campenhout A, Deschepper E, Van den Broeck C, Desloovere K. Progressive resistance training for children with cerebral palsy: A randomized controlled trial evaluating the effects on muscle strength and morphology. Front Physiol. 2022 Oct 4;13:911162. doi: 10.3389/fphys.2022.911162. eCollection 2022. PMID 36267577
- [Result] Verreydt I, Vandekerckhove I, Stoop E, Peeters N, van Tittelboom V, Van de Walle P, Van den Hauwe M, Goemans N, De Waele L, Van Campenhout A, Hanssen B, Desloovere K. Instrumented strength assessment in typically developing children and children with a neural or neuromuscular disorder: A reliability, validity and responsiveness study. Front Physiol. 2022 Oct 19;13:855222. doi: 10.3389/fphys.2022.855222. eCollection 2022. PMID 36338500
- [Result] Vandekerckhove I, Hanssen B, Peeters N, Dewit T, De Beukelaer N, Van den Hauwe M, De Waele L, Van Campenhout A, De Groote F, Desloovere K. Anthropometric-related percentile curves for muscle size and strength of lower limb muscles of typically developing children. J Anat. 2025 Aug;247(2):348-362. doi: 10.1111/joa.14241. Epub 2025 Mar 17. PMID 40098309

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All children aged 5-11 years old were extracted from the database of the CP reference center Leuven (n=342) and screened based on gross motor function classification system level and type of CP. The appointments at the hospital were checked monthly to further screen potential participants (±10% eligible every month, part of the n=342). Additionally, pediatric physiotherapists at private practices and special needs schools were consulted for potential participants (n=6 not followed in Leuven).
Groups:
- Intervention Group: During 12 weeks, children receive 3-4 sessions of progressive strength training per week (on top of the usual care.) All children will be provided with an individualized training program and supporting equipment. One or 2 sessions per week will be performed under the supervision of the physical therapist, whilst the remaining sessions will be conducted at home. The principal investigator and training programs closely monitor progression are adjusted if necessary.
  Progressive strength training: Progressive Supervised Home-based Strength Training
Period: Overall Study
Arm/Group | Intervention Group | Waitlist-control Group
Started | 27 | 22
Completed | 19 | 19
Not Completed | 8 | 3
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Did not receive intervention (inability to cooperate with assessment or cancellation due to Covid) | 2 | 0

BASELINE CHARACTERISTICS:
Population: For parameters that could be assessed per leg, both legs of bilaterally affected participants were included and only the affected leg of unilaterally affected participants.
Units Other Than Participants: Legs
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Waitlist-control Group | Total
Number analyzed (Participants) | 26 | 22 | 48
Number analyzed (Legs) | 41 | 36 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 22 | 48
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.3 (2.0) | 8.5 (2.1) | 8.4 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 14 | 16 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 26 | 22 | 48
Involvement [Count of Participants; unit: Participants]
  Unilateral | 11 | 8 | 19
  Bilateral | 15 | 14 | 29
Gross motor function classification system [Count of Participants; unit: Participants] — The Gross Motor Function Classification System (GMFCS) is a five-level scale used to describe the movement abilities of children and youth with cerebral palsy, ranging from Level I (most independent) to Level V (most limited mobility). Children with levels I to III were included in this study, indicating children who are ambulatory.
  Participants
    Level I | 17 | 14 | 31
    Level II | 5 | 5 | 10
    Level III | 4 | 3 | 7
Weight [Mean (Standard Deviation); unit: kilogram] | 27.7 (8.1) | 28.3 (7.1) | 28.0 (7.6)
Height [Mean (Standard Deviation); unit: centimeter] | 127.3 (14.0) | 128.6 (11.2) | 127.9 (12.7)
Fibula length [Mean (Standard Deviation); unit: millimeter] | 27.7 (3.6) | 27.8 (3.5) | 27.7 (3.5)
Selective control assessment of the lower extremity (score out of 10) [Mean (Standard Deviation); unit: units on a scale] — The Selective Control Assessment of the Lower Extremity (SCALE) is a clinical tool used to measure how well someone with cerebral palsy can intentionally move individual joints in their legs without unwanted movement in other parts. The SCALE consists of 5 subtests (hip, knee, ankle, subtalar joint and toes) each scored a 0, 1 or 2. The total score for one leg ranges therefor from 0 to 10.
  units on a scale | 7.0 (2.1) | 7.1 (2.6) | 7.0 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Muscle Size Parameter
Description: Estimation of muscle volume by 3D freehand ultrasonography.
Time Frame: baseline, post-intervention (12-weeks)
Population: There were some missing data due to 3DfUS reconstructions that could not be (fully) analyzed because of technical errors, isometric and functional strength tests that could not be assessed due to inability of the participant and missing anthropometric information.
Measure: Mean (95% Confidence Interval); unit: milliliters
Units Other Than Participants: Affected legs
Arm/Group | Intervention Group | Waitlist-control Group
Number analyzed (Participants) | 26 | 22
Number analyzed (Affected legs) | 41 | 36
milliliters
  Muscle volume - rectus femoris: number analyzed (Affected legs) | 41 | 35
  Muscle volume - rectus femoris | 3.7 [1.9 to 5.5] | 1.6 [-0.1 to 3.4]
  Muscle volume - semitendinosis: number analyzed (Affected legs) | 38 | 31
  Muscle volume - semitendinosis | 1.4 [-0.5 to 3.3] | 0.1 [-1.8 to 2.0]
  Muscle volume - medial gastrocnemius | 2.0 [0.9 to 3.1] | 0.5 [-0.5 to 1.6]
Statistical Analysis 1: Comparison: Intervention Group vs Waitlist-control Group; Test type: Superiority; p < 0.01, Mixed Models Analysis — The α-level was adjusted to p ≤ 0.01 since multiple parameters were evaluated for most research questions, with a maximum of 5 parameters (functional strength)

2. Primary Outcome: Change in Muscle Length
Description: Estimation of muscle length parameters by 3D freehand ultrasonography from origo to muscle tendon junction.
Time Frame: baseline, post-intervention (12-weeks)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: millimeters
Units Other Than Participants: Affected legs
Arm/Group | Intervention Group | Waitlist-control Group
Number analyzed (Participants) | 26 | 22
Number analyzed (Affected legs) | 41 | 36
millimeters
  Muscle length - rectus femoris: number analyzed (Affected legs) | 40 | 33
  Muscle length - rectus femoris | 3.9 [0.0 to 7.7] | 5.5 [1.8 to 9.3]
  Muscle length - semitendinosis: number analyzed (Affected legs) | 35 | 31
  Muscle length - semitendinosis | 3.2 [-1.3 to 7.7] | 3.0 [-1.6 to 7.5]
  Muscle length - medial gastrocnemius: number analyzed (Affected legs) | 41 | 34
  Muscle length - medial gastrocnemius | 3.5 [1.4 to 5.6] | 2.4 [0.3 to 4.4]
Statistical Analysis 1: Comparison: Intervention Group vs Waitlist-control Group; Test type: Superiority; p < 0.01, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Change in Echogenicity Intensity
Description: Estimation of echogenicity intensity by 3D freehand ultrasonography on an 8-bit greyscale (256 values ranging from 0 to 255). Echogenicity intensity was defined over the whole muscle volume.
  Echogenicity intensity refers to the brightness of a muscle seen on the ultrasound image, which reflects how much sound is being bounced back (or "echoed") by the tissue. Higher echo-intensity (i.e., higher values) often indicates increased fat or fibrous tissue within the muscle and is therefore seen as a worse outcome. Whereas low echo-intensity (i.e., lower values) indicate less non-muscular tissue in the muscle, therefor higher quality and a better outcome.
Time Frame: baseline, post-intervention (12-weeks)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: arbitrary units
Units Other Than Participants: legs
Arm/Group | Intervention Group | Waitlist-control Group
Number analyzed (Participants) | 26 | 22
Number analyzed (legs) | 41 | 36
arbitrary units
  Echo-intensity - rectus femoris: number analyzed (legs) | 41 | 35
  Echo-intensity - rectus femoris | -0.3 [-4.6 to 3.9] | -0.1 [-4.2 to 4.1]
  Echo-intensity - semitendinosus: number analyzed (legs) | 38 | 31
  Echo-intensity - semitendinosus | 3.8 [-1.1 to 8.7] | 3.2 [-1.9 to 8.3]
  Echo-intensity - medial gastrocnemius: number analyzed (legs) | 41 | 35
  Echo-intensity - medial gastrocnemius | 0.2 [-3.0 to 2.4] | 1.8 [-1.4 to 4.9]
Statistical Analysis 1: Comparison: Intervention Group vs Waitlist-control Group; Test type: Superiority; p < 0.01, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

4. Primary Outcome: Change in Isometric Muscle Strength
Description: Evaluation of isometric muscle strength by Instrumented Weakness Assessment.
Time Frame: baseline, post-intervention (12-weeks)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Newton meters
Units Other Than Participants: legs
Arm/Group | Intervention Group | Waitlist-control Group
Number analyzed (Participants) | 26 | 22
Number analyzed (legs) | 41 | 36
Newton meters
  Knee extension strength: number analyzed (legs) | 39 | 36
  Knee extension strength | 2.5 [0.8 to 4.2] | -0.4 [-2.1 to 1.2]
  Knee flexion strength: number analyzed (legs) | 39 | 36
  Knee flexion strength | 6.0 [3.3 to 8.7] | 0.8 [-1.9 to 3.4]
  Plantar flexion strength: number analyzed (legs) | 39 | 35
  Plantar flexion strength | 3.6 [2.2 to 5.0] | 1.1 [-0.3 to 2.5]
Statistical Analysis 1: Comparison: Intervention Group vs Waitlist-control Group; Test type: Superiority; p < 0.01, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

5. Primary Outcome: Change in Functional Muscle Strength - Muscle Endurance
Description: Evaluation of functional muscle strength by 30-sec maximum repetition tests of the Adapted Functional Strength measure.
  For unilateral exercises (lateral step-up and unilateral heel raise) all affected legs were assessed.
Time Frame: baseline, post-intervention (12-weeks)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: repetitions
Units Other Than Participants: legs
Arm/Group | Intervention Group | Waitlist-control Group
Number analyzed (Participants) | 26 | 22
Number analyzed (legs) | 41 | 36
repetitions
  Sit-to-stand: number analyzed (Participants) | 25 | 21
  Sit-to-stand: number analyzed (legs) | 25 | 21
  Sit-to-stand | 2.7 [1.2 to 4.1] | 0.3 [-1.3 to 1.9]
  Lateral step-up: number analyzed (legs) | 38 | 34
  Lateral step-up | 2.7 [1.4 to 3.9] | 1.1 [-0.2 to 2.3]
  Bilateral heel raise: number analyzed (Participants) | 22 | 22
  Bilateral heel raise: number analyzed (legs) | 22 | 22
  Bilateral heel raise | 4.5 [1.9 to 7.1] | 3.6 [1.1 to 6.0]
  Unilateral heel raise: number analyzed (legs) | 27 | 27
  Unilateral heel raise | 9.1 [5.7 to 12.4] | -1.5 [-4.7 to 1.7]
Statistical Analysis 1: Comparison: Intervention Group vs Waitlist-control Group; Test type: Superiority; p < 0.01, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change in Gross Motor Function
Description: Evaluation of gross motor function by the Gross Motor Function Measure (GMFM) item set. The GMFM is a standardized observational tool used to assess motor function in children with cerebral palsy by evaluating specific physical tasks across five areas: lying & rolling, sitting, crawling & kneeling, standing, and walking/running/jumping. Each item is scored on a 4-point scale: 0 (does not initiate), 1 (initiates but completes less than 10%), 2 (partially completes, 10% to less than 100%), and 3 (fully completes). Higher scores indicate better gross motor function, with a maximum of 66.
Time Frame: baseline, post-intervention (12 weeks)
Population: There were some missing data due to 3DfUS reconstructions that could not be (fully) analyzed because of technical errors, isometric and functional strength tests that could not be assessed due to inability of the participant.
  and missing anthropometric information.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Waitlist-control Group
Number analyzed (Participants) | 26 | 21
score on a scale | 0.7 [-0.6 to 2.1] | 0.3 [-1.1 to 1.8]
Statistical Analysis 1: Comparison: Intervention Group vs Waitlist-control Group; Test type: Superiority; p < 0.01, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

7. Other Pre Specified Outcome: Change in Quality of Life
Description: Evaluation of quality of life by the CP Quality of Life (CP QOL-Child) questionnaire for children. This questionnaire evaluates quality of life over various domains on a 1-9 scale. A higher score indicates more happiness.
Time Frame: baseline, post-intervention (12 weeks)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Functionality
Description: The level of functionality and activity is assessed by the Gillette Functional Assessment questionnaire. This parent-reported questionnaire consists of 22 items (0 low function - 10 high function).
Time Frame: baseline, post-intervention (12 weeks)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Patient Reported Physical Function
Description: The perceived level of physical functioning is assessed by the Activities Scale for Kids
Time Frame: Baseline, post-intervention (12 weeks)
Reporting Status: Not Posted

10. Primary Outcome: Change in Functional Muscle Strength - Maximum Jumping Distance
Description: Evaluation of standing long jump by the Adapted Functional Strength measure.
Time Frame: baseline, post-intervention (12-weeks)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: distance in centimer
Arm/Group | Intervention Group | Waitlist-control Group
Number analyzed (Participants) | 19 | 16
distance in centimer | 5.8 [-0.2 to 11.8] | 2.7 [-2.8 to 8.3]
Statistical Analysis 1: Comparison: Intervention Group vs Waitlist-control Group; Test type: Superiority; p < 0.01, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

11. Secondary Outcome: Change in Walking Capacity
Description: Evaluation of walking capacity by assessing the distance covered during the 1-minute walking test
Time Frame: baseline, post-intervention (12 weeks)
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: distance in meters
Arm/Group | Intervention Group | Waitlist-control Group
Number analyzed (Participants) | 22 | 21
distance in meters | 5.6 [0.9 to 10.4] | 3.6 [-1.0 to 8.1]
Statistical Analysis 1: Comparison: Intervention Group vs Waitlist-control Group; Test type: Superiority; p < 0.01, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Intervention Group | Waitlist-control Group
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/22
Other Adverse Events (participants affected / at risk) | 10/26 | 0/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=26) | Waitlist-control Group (N=22)
muscle cramp or pain, joint pain and general discomfort from the weighted vest (Musculoskeletal and connective tissue disorders) | 10 (10) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT03863197/Prot_SAP_000.pdf